## Patients consent form cover page

Official study title: Multicenter registry to study the characteristic and outcomes of Jordanian Heart Failure patients
The Jordanian Heart Failure Registry ( JoHFR)
NCT04829591

The actual document and approval date 30/3/2021 The updated document date 17/4/2021

## Consent form

| I the undersigned | |
|-------------------|------|
| | <br> |

Consent to the investigators in the heart failure Jordanian study to share information regarding my medical background and current medical illnesses for the sole purpose of including it in this registry.

I do understand that my identity and my private information will not be shared with the investigators for any reason.

And I do understand that this is a non-intervention registry study which does not entitle the investigators to give me any specific, not approved medication or subject me to any investigation which are not medically needed.

Signature.